CLINICAL TRIAL: NCT03731676
Title: Outcomes of Rotating Platform Versus Mobile Bearing Total Knee Arthroplasty
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: William Hopkinson (Other)
Responsible Party: Sponsor-Investigator, William Hopkinson, Professor, Vice Chairman of Orthopaedic Surgery and Rehabilitation, Loyola University
Organization: Loyola University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 11119
Record Dates: First submitted 2018-10-16; First posted 2018-11-06 (Actual); Last update posted 2021-04-19 (Actual); Status verified 2021-04

CONDITIONS: Total Knee Arthroplasty

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Rotating platform total knee arthroplasty (Active Comparator): These patients were randomly assigned to receive a rotating platform total knee arthroplasty.
  Interventions: Device: Rotating platform total knee arthroplasty
- Fixed bearing total knee arthroplasty (Active Comparator): These patients were randomly assigned to receive a fixed bearing total knee arthroplasty.
  Interventions: Device: Fixed bearing total knee arthroplasty

INTERVENTIONS:
Device: Fixed bearing total knee arthroplasty — Fixed bearing total knee arthroplasty
  Arms: Fixed bearing total knee arthroplasty
Device: Rotating platform total knee arthroplasty — Rotating platform total knee arthroplasty
  Arms: Rotating platform total knee arthroplasty

SUMMARY:
Patients were randomly assigned to a fixed bearing or rotating platform of two prostheses. A subsequent study (the one retrospectively registering the original study) asked these patients a series of questions from published questionnaires to assess long term outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Osteoarthritis
2. Rheumatoid or other inflammatory arthritis
3. Post-traumatic arthritis
4. Juvenile rheumatoid arthritis
5. Avascular necrosis

Exclusion Criteria:

1. History of recent/active joint sepsis
2. Charcot neuropathy
3. Psycho-social disorders that would limit rehabilitation
4. Metabolic disorders of calcified tissues, such as Paget's disease
5. Joint replacement due to autoimmune disorders
6. Skeletal immaturity
7. Ligamentous laxity requiring a constrained prosthesis

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2000-12-01 (Actual); Primary Completion 2001-12-31 (Actual); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Functional Status over time | Pre-operative, Post-operative Week 6, Month 3, Month 6, Year 1, Year 2, Year 5, Year 10, Year 12, Year 15 and Year 20.
  Knee Society Clinical Rating Scale
Change in Osteoarthritis Status over time | Pre-operative, Post-operative Week 6, Month 3, Month 6, Year 1, Year 2, Year 5, Year 10, Year 12, Year 15 and Year 20.
  Western Ontario and McMaster University Osteoarthritis Index (WOMAC)- A 24 item questionnaire to assess pain, stiffness, and physical function in patients with hip or knee osteoarthritis divided into 3 subscales: Pain (5 items), Stiffness (2 items), Physical function (17 items)
Change in Overall Health Status over time | Pre-operative, Post-operative Week 6, Month 3, Month 6, Year 1, Year 2, Year 5, Year 10, Year 12, Year 15 and Year 20.
  Medical Outcomes Study Short Form -36 Health Survey (SF-36)- A 36 item questionnaire to assess overall health.

SECONDARY OUTCOMES:
Change in Satisfaction of Knee over time | Pre-operative, Post-operative Week 6, Month 3, Month 6, Year 1, Year 2, Year 5, Year 10, Year 12, Year 15 and Year 20.
  4-point Likert scale used to assess satisfaction with knee Scale-1. Extremely satisfied 2. Satisfied 3. Unsatisfied 4. Extremely unsatisfied

CONTACTS AND LOCATIONS:
Locations (1):
- Dr. William Hopkinson, Maywood, Illinois, United States

IPD SHARING:
Plan to Share IPD: No
Results in a general basis via a manuscript. No individual data.